CLINICAL TRIAL: NCT06969508
Title: The Relationship Between Core Stabilization Exercises and Paraspinal Muscle Thickness in Chronic Low Back Pain
Brief Title: Effect Of Paraspinal Muscle Thickness On The Benefit Of Core Stabilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Collaborators: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Mucahit Atasoy, MD, Asst. Prof. MD, Medipol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KAEK-11
Record Dates: First submitted 2025-04-24; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Back Pain Lower Back Chronic; Lumbar Disc Degenerative Disease
Keywords: Paraspinal Muscles; exercise; Low Back Pain
MeSH Terms: conditions — Intervertebral Disc Degeneration; Motor Activity; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Lumbar disc herniation (Experimental): This study involved a single cohort of participants who had been diagnosed with chronic non-specific low back pain. All participants had lumbar MRI scans performed at least 6 months prior to enrollment to confirm the absence of severe pathology requiring surgical intervention. This cohort received a 6-month exercise program specifically designed to target and strengthen the core stabilizing muscles of the spine, including the multifidus, transversus abdominis, and pelvic floor muscles. The exercise program was provided to participants through videotaped instructions demonstrating the correct form and technique for each exercise. Participants were instructed to perform these exercises at home, following the provided video guidance. At the beginning of the study, the thickness of their paraspinal muscles (specifically the multifidus) was measured. The study assessed the changes in their pain levels and functional status over the 6-month period, with measurements taken at baseline, 3 mon
  Interventions: Other: core stabilitation exercises

INTERVENTIONS:
Other: core stabilitation exercises — The core stabilization exercise program aimed to strengthen deep spinal muscles: transversus abdominis (abdominal bracing), multifidus (segmental stability), and pelvic floor muscles (pelvic support). Participants received videotaped instructions for performing these exercises at home regularly for 6 months, with a gradual increase in difficulty.

SUMMARY:
This study investigates whether the effects of core muscle strengthening exercises on chronic low back pain and deep back muscle (multifidus) thickness differ in patients with different baseline muscle thicknesses. Pain levels will be measured before and after a 6-month exercise program in patients with different baseline muscle thicknesses. The aim is to determine whether the exercises are more or less effective depending on the baseline condition of these muscles. Understanding this may help personalize exercise treatments for chronic low back pain based on individual muscle characteristics.

DETAILED DESCRIPTION:
This prospective, randomized study will investigate if the initial thickness of deep back muscles (multifidus and erector spinae), measured via existing lumbar MRI scans, influences the effectiveness of a 6-month core stabilization exercise program for chronic low back pain. Participants aged 20-60 with chronic low back pain (over 3 months) and a recent lumbar MRI will be recruited from Çam Sakura City Hospital. Individuals with prior spinal surgery, previous physical therapy, neurological or cardiorespiratory issues, or osteoporosis will be excluded.

At baseline, muscle thickness at the L4/L5 level will be measured. Participants will receive a home-based core stabilization exercise program. Pain and function will be assessed using VAS, Oswestry Disability Index, and SPI at baseline, 3, and 6 months. The study aims to determine if patients with different baseline muscle thicknesses show varying degrees of improvement in pain and function following the exercise program. Correlation and regression analyses will explore the relationship between initial muscle thickness and changes in outcome measures. The findings may help personalize exercise treatments for chronic low back pain based on individual muscle characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic low back pain: Participants had to have experienced low back pain for at least 3 months,
* Lumbar MRI findings without severe pathology requiring surgical intervention: Participants' lumbar MRI scans, performed at least 6 months prior to enrollment, had to show evidence of low back pain-related findings but exclude conditions necessitating surgical treatment.
* Willingness to participate in the study and provide informed consent: Participants had to voluntarily agree to take part in the research and provide their written informed consent.

Exclusion Criteria:

* History of prior spinal surgery: Individuals who had undergone any previous surgical procedures on their spine were not eligible.

Diagnosis of a neurological or rheumatological disease: Participants with pre-existing neurological conditions (e.g., radiculopathy with significant motor deficit) or rheumatological diseases (e.g., ankylosing spondylitis) were excluded.

* Cardiovascular or pulmonary comorbidities: Individuals with significant heart or lung conditions that could affect their ability to participate in the exercise program were excluded.
* Osteoporosis or osteoporotic vertebral fracture: Participants with known osteoporosis or a history of vertebral fracture due to osteoporosis were not eligible.
* Currently receiving physical therapy modalities or oral/algologic injections for low back pain: Individuals already undergoing other active treatments for their low back pain were excluded to avoid confounding the results.
* Unwillingness to participate in the study or provide informed consent: Individuals who did not want to take part in the research or were unable to provide their written informed consent were excluded.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
VAS score | Baseline, 3 months, 6 months
  Pain intensity was measured using a Visual Analog Scale (VAS) ranging from 0 to 10 centimeters (cm). Zero (0 cm) was equivalent to "no pain," and 10 centimeters (10 cm) indicated the "worst imaginable pain." Changes in VAS scores were assessed at 3 and 6 months to determine the effect of the exercise program on pain levels.
Brief Pain İnventory- Short Form | Baseline, 3 months, 6 months
  Pain intensity was assessed using the Brief Pain Inventory - Short Form (BPI-SF). Participants were asked to rate their pain at its worst, least, average, and current level on a scale ranging from 0 to 10, where 0 indicated "no pain" and 10 indicated "pain as bad as you can imagine." Changes in these pain intensity scores were assessed at 3 and 6 months to determine the effect of the exercise program on different dimensions of pain experience.
  Pain interference was assessed using the Brief Pain Inventory - Short Form (BPI-SF). Participants were asked to rate how much their pain interfered with seven aspects of their daily life (general activity, mood, walking ability, normal work, sleep, enjoyment of life, and relations with other people) on a scale ranging from 0 to 10, where 0 indicated "does not interfere" and 10 indicated "completely interferes." Changes in these pain interference scores (either individual item scores or a composite score calculated as the mean of the seven items)
Oswestry Disability Index (ODI) | Baseline, 3 months, 6 months
  Functional disability was assessed using the Oswestry Disability Index (ODI), a ten-section questionnaire. Each section is scored from 0 (no disability) to 5 (severe disability). The total score, converted to a percentage ranging from 0% (no disability) to 100% (most severe disability), reflects the level of functional limitation due to back pain. Changes in the total ODI score were assessed at 3 and 6 months to evaluate the impact of the exercise program on functional disability.
Baseline thickness of the paraspinal muscles | Baseline
  The thickness of the paraspinal muscles, specifically the multifidus muscle at the L4-L5 vertebral level, was measured on both the right and left sides at the beginning of the study using Magnetic Resonance Imaging (MRI). These measurements represent the initial size of the multifidus muscle in the participants prior to the start of the exercise program.

SECONDARY OUTCOMES:
Correlation between baseline thickness of the paraspinal muscles as measured by MRI and the change in pain intensity | Baseline, 6 months
  This outcome measure will assess the statistical relationship between the initial thickness of the multifidus muscle (measured on both the right and left sides at baseline via MRI) and the change in pain intensity as reported on the Visual Analog Scale (VAS) from baseline to the 6-month follow-up. The correlation coefficient will indicate the strength and direction of this relationship.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Çam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No. While we are open to sharing individual participant data (IPD) with other researchers upon reasonable request, there is no specific platform or repository designated for making this data publicly available. Interested researchers should contact the corresponding author to inquire about data sharing, and any data transfer will be subject to ethical considerations and data sharing agreements.

REFERENCES:
- [Background] Wong AYL, Parent EC, Funabashi M, Stanton TR, Kawchuk GN. Do various baseline characteristics of transversus abdominis and lumbar multifidus predict clinical outcomes in nonspecific low back pain? A systematic review. Pain. 2013 Dec;154(12):2589-2602. doi: 10.1016/j.pain.2013.07.010. Epub 2013 Jul 16. PMID 23867731
- [Background] Li Y, Yan L, Hou L, Zhang X, Zhao H, Yan C, Li X, Li Y, Chen X, Ding X. Exercise intervention for patients with chronic low back pain: a systematic review and network meta-analysis. Front Public Health. 2023 Nov 17;11:1155225. doi: 10.3389/fpubh.2023.1155225. eCollection 2023. PMID 38035307
- [Background] Wang XQ, Zheng JJ, Yu ZW, Bi X, Lou SJ, Liu J, Cai B, Hua YH, Wu M, Wei ML, Shen HM, Chen Y, Pan YJ, Xu GH, Chen PJ. A meta-analysis of core stability exercise versus general exercise for chronic low back pain. PLoS One. 2012;7(12):e52082. doi: 10.1371/journal.pone.0052082. Epub 2012 Dec 17. PMID 23284879